CLINICAL TRIAL: NCT03284476
Title: A Prospective Cohort of Patients Hospitalized in West French Intensive Care Units for Peritonitis Surgically Treated
Brief Title: Post Surgically Treated Peritonitis Complications
Status: Withdrawn | Type: Observational
Why Stopped: No inclusion
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC12_0207 doublon
Record Dates: First submitted 2017-09-14; First posted 2017-09-15 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Peritonitis
Keywords: Nosocomial Peritonitis; Community-acquired Peritonitis; Post-operative Peritonitis
MeSH Terms: conditions — Peritonitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICU patients: Collection of medical data of Patients with peritonitis (nosocomial or community-acquired) or Patients with post-operative peritonitis
  Interventions: Other: Collection of medical data from ICU patients

INTERVENTIONS:
Other: Collection of medical data from ICU patients — Medical data collected on a electronic secured data base

SUMMARY:
The purpose of this observational study is to investigate the management and the complications associated wtih surgically treated peritonitis.

Data will be analysed to answer pre-defined scientific projects and to improve management of these conditions.

DETAILED DESCRIPTION:
Anonymous data will be collected by study coordinators in a secured e-database. Cross audit will be performed to check data.

ELIGIBILITY:
Inclusion Criteria:

* Nosocomial surgically treated Peritonitis
* Or Community-Acquired surgically treated Peritonitis
* Or Post-operative surgically treated Peritonitis

Exclusion Criteria:

* Consent withdrawal

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized in ICU for peritonitis surgically treated
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-04 (Estimated); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
In ICU stay main complications | Within the first 28 days after ICU admission date
  Nosocomial Infections (epidemiology, risk factors, antibiotic susceptibility of pathogens) Organ failures (incidence, risk factors)

SECONDARY OUTCOMES:
Duration of mechanical ventilation | In ICU (up to 90 days)
ICU length of stay | In ICU (up to 90 days)

OTHER OUTCOMES:
Death | In ICU (up to 90 days)

CONTACTS AND LOCATIONS:
Overall Officials: Karim Asehnoune, MD, PhD, Study Chair — Non Affiliated
Locations (5):
- France (5):
  - Angers University Hospital, Angers
  - Nantes University Hospital, Nantes
  - Poitiers University Hospital, Poitiers
  - Rennes University Hospital, Rennes
  - Tours University Hospital, Tours